CLINICAL TRIAL: NCT01639950
Title: Validation of the English Version of the Pain Interference Index and the Pain Rating Scale in Children, Adolescents, and Adults With Chronic Illness and Their Parents
Brief Title: Validating Pain Scales in Children and Young Adults
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 120160; 12-C-0160
Record Dates: First submitted 2012-07-11; First posted 2012-07-13 (Estimated); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Sickle Cell Disease; Solid Tumor; Leukemia; Neurofibromatosis
Keywords: Self-Report; Survey Scale; Validate; Pain Severity; Reliability; Natural History
MeSH Terms: conditions — Anemia, Sickle Cell; Leukemia; Neurofibromatoses; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Adults Group 1: Adults patients with cancer or neurofibromatosis 1 (NF1)
- Adults Group 2: Adults with sickle cell disease (SCD)
- Children: Children with with neurofibromatosis 1 (NF1), genetic tumor predisposition syndromes (GTPS), malignant solid tumor, or leukemia. -closed
- Parents: Parents of children with with neurofibromatosis 1 (NF1), genetic tumor predisposition syndromes (GTPS), malignant solid tumor, or leukemia. -closed

SUMMARY:
Background:

- Assessing pain levels is important to improve treatments for different illnesses. Most pain rating scales are used to determine pain levels in adults. Pain is also a common symptom among children who have cancer. Those who have genetic conditions that may lead to cancer may also have pain symptoms. However, the pain scales used for adults have not been fully tested in children and young adults. As a result, they may not be as accurate. Researchers want to test pain rating scales in children and young adults who have cancer and genetic conditions that can lead to cancer.

Objectives:

- To study the effectiveness of pain rating scales given to children and adults with Sickle Cell Disease (SCD),cancer, and related genetic conditions.

Eligibility:

- Adults 18 and 34 years of age and older who have SCD, cancer, or other genetic conditions that can lead to cancer.

Design:

* Participants with SCD, cancer or related genetic conditions will fill out four questionnaires. These questionnaires will ask about pain levels and how much pain interferes with daily life.
* Pain treatments will not be provided as part of this study.

DETAILED DESCRIPTION:
Background:

Pain is a common symptom among children with a variety of medical illnesses. Currently, a number of rating scales are used to assess pain interference and pain severity in adults. However, relatively few measures assessing these variables have been validated for use with children and adolescents, and existing tools have limitations.

Objectives:

The primary objective is to validate the self-report and parent versions of the Pain Interference Index (PII) and the Pain Rating Scale (PRS) by comparison with previously validated measures of pain interference (Modified Brief Pain Inventory) and pain severity (Faces Pain Scale - Revised) in the following populations:

-Children, adolescents, and young adults ages 8 to 25 years with chronic pain related to cancer, Neurofibromas type 1 (NF1), genetic tumor predisposition syndromes (GTPS), a solid tumor (including but not limited to sarcoma, neuroblastoma, or melanoma), or

leukemia and their parent(s) or guardians. (COMPLETED)

Adults > =18 years of age with cancer, NF1, Sickle Cell Disease (SCD)

Eligibility:

* >= 18 years of age
* Diagnosis of cancer, NF1, SCD
* Enrolled on a clinical trial or natural history study at the NIH Clinical Center

Design:

* Eligible participants will be asked to respond one time to the PII and the PRS, as well as the Modified Brief Pain Inventory and Faces Pain Scale - reviewed during a scheduled clinic visit for their primary protocol, over video conferencing, or while inpatient.
* Demographic (gender and age, parent gender (if applicable) and medical (diagnosis, date of diagnosis, pain medication) data will be collected from review of the participants medical record.
* A subset of evaluable participants with SCD will be asked to repeat the PII after

approximately 1 month to assess test-retest reliability in this tool.

* Parents of pediatric participants were asked to complete the Parent version of the PII and the Parent PRS. Correlations between patient participant and parent participant questionnaire results for participants with solid tumor, NF1, GTPS, and leukemia will be correlated to establish validity and reliability of the PII and PRS. (COMPLETE)
* Also, results from mother and father reports will be correlated to assess inter-rater

reliability. (COMPLETE)

-Data from 12 participants ages 6 and 7 years was collected to determine the feasibility of the forms in this younger age group. (COMPLETE)

ELIGIBILITY:
* IINCLUSION CRITERIA:
* Participants must have a cytologically confirmed cancer, SCD, or meet the diagnostic criteria for NF1 documented in the medical record according to the primary treatment or natural history protocol. Participants must be at least one month post-diagnosis.
* Age >= 18
* Participants who complete the pain interference measure (the Pain Interference Index PII) and the pain severity tool (Pain Rating Scale PRS) once but who miss their Time 2 evaluation, are eligible to enroll a second time to complete the measures again in order to participate in the test-retest reliability assessment.
* Ability to read and/or understand English

EXCLUSION CRITERIA:

Participants may be excluded from this study if in the judgment of the Principal or Associate Investigator, the subject is too ill, or subject s cognitive ability would compromise their ability to participate in study related procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Children, adolescents, and young adults ages 6 to 25 years with chronic pain related to cancer, Neurofibromas type 1 (NF1), genetic tumor predisposition syndromes (GTPS), a solid tumor (including but not limited to sarcoma, neuroblastoma, or melanoma), or leukemia and their parent(s) or guardians. (COMPLETED) Adults >/= 18 years of age with cancer, NF1, Sickle Cell Disease (SCD)
Sampling Method: Non-Probability Sample
Enrollment: 252 (Actual)
Dates: Start 2012-08-06 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-06-28 (Actual)

PRIMARY OUTCOMES:
Feasability | One time
  To validate the Pain Interference Index and the Pain Rating Scale by comparison with previously validated measures

SECONDARY OUTCOMES:
Validation | One month
  To establish the reliability (internal consistency and inter-rater) of the PII and PRS
Feasability | One time
  To establish normative data for the PII and PRS.
Feasability | One time
  To gather preliminary data on the feasibility of using the PII and PRS with children ages 6 and 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Staci M Peron, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
.All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- [Background] Fayers PM, Hjermstad MJ, Klepstad P, Loge JH, Caraceni A, Hanks GW, Borchgrevink P, Kaasa S; European Palliative Care Research Collaborative (EPCRC). The dimensionality of pain: palliative care and chronic pain patients differ in their reports of pain intensity and pain interference. Pain. 2011 Jul;152(7):1608-1620. doi: 10.1016/j.pain.2011.02.052. Epub 2011 Apr 1. PMID 21458921
- [Background] Hjermstad MJ, Fayers PM, Haugen DF, Caraceni A, Hanks GW, Loge JH, Fainsinger R, Aass N, Kaasa S; European Palliative Care Research Collaborative (EPCRC). Studies comparing Numerical Rating Scales, Verbal Rating Scales, and Visual Analogue Scales for assessment of pain intensity in adults: a systematic literature review. J Pain Symptom Manage. 2011 Jun;41(6):1073-93. doi: 10.1016/j.jpainsymman.2010.08.016. PMID 21621130
- [Background] Engel JM, Jensen MP, Ciol MA, Bolen GM. The development and preliminary validation of the pediatric survey of pain attitudes. Am J Phys Med Rehabil. 2012 Feb;91(2):114-21. doi: 10.1097/PHM.0b013e318238a074. PMID 22019973
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2012-C-0160.html